CLINICAL TRIAL: NCT05951283
Title: A Longitudinal, Single Centre Study to Assess the Effects of Artificial Pancreas-related Changes in Diabetic Neuropathy
Brief Title: Quantifying Artificial Pancreas-related Changes in Diabetic Neuropathy
Acronym: QUANT-AP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B01841
Record Dates: First submitted 2023-03-16; First posted 2023-07-19 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Complications; Diabetes Mellitus, Type 1; Diabetic Neuropathies
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus, Type 1; Diabetic Neuropathies; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MDI (No Intervention): All participants will have:
  Continuous Glucose Monitoring Neuropathy Assessments and Pain Questionnaires ACR, Blood Tests
- Artificial Pancreas - Closed Loop (Active Comparator): All participants will have:
  Continuous Glucose Monitoring Neuropathy Assessments and Pain Questionnaires ACR, Blood Tests
  Interventions: Device: Hybrid Closed Loop Insulin Pump

INTERVENTIONS:
Device: Hybrid Closed Loop Insulin Pump — As above
  Arms: Artificial Pancreas - Closed Loop

SUMMARY:
A complication of diabetes mellitus is damage to nerves called neuropathy. There are several mechanisms involved that will lead to the development of neuropathy. Neuropathy can lead to foot ulcers, infections and amputations. Patients with neuropathy may also experience pain, which can be difficult to control and the medications are limited by side effects. Despite this there are no approved treatments to reverse the progression of neuropathy and the management of patients is focused on controlling blood glucose and other metabolic factors to prevent neuropathy and its symptoms from getting worse.

Patients with type 1 diabetes are prescribed multiple daily injections (MDI) of insulin to manage their glucose control. However, insulin pump therapy and, more recently, automated insulin delivery (AID) or the Artificial Pancreas can be used as the insulin delivery method for patients with type 1 diabetes mellitus. Manchester Diabetes Centre is the first adult diabetes centre in Europe to pioneer and use a commercially-approved AID in clinical practice.

Insulin pump therapy and AID have the advantage of being able to provide insulin at variable doses, which is closer to the natural process occurring within an individual without diabetes. Both are currently considered to be the most physiological method of insulin delivery and have been shown to improve glycaemic control, quality of life (QOL) and reduce the risk of hypoglycaemia (low blood glucose level). The investigators have previously shown in a small group of people that use of an insulin pump therapy may improve symptoms of painful neuropathy via a more stable glucose profile. The peaks and drops in insulin may make neuropathy worse.

In this study the investigators aim to investigate the use of insulin pump therapy and AID in their effect on neuropathy. This will be in comparison to a control group of patients on MDI. The investigatorsbwill use a variety of neuropathy measures and symptom questionnaires to assess structural and functional neuropathy status. The investigators hypothesise that those patients receiving the newer technologies will demonstrate an improvement in symptoms and nerve regeneration.

This finding would have a significant impact for patients as it would provide evidence to suggest that those patients with neuropathy should be put onto an insulin pump or AID to improve neuropathy and its symptoms. As these are treatments that are already available on the NHS to patients satisfying specific criteria this study aims to show benefit in this cohort of patients which can be implemented immediately in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Type 1 diabetes aged 18-70 who falls into either of these three categories and has the ability to read and comprehend English:

Starting Artificial Pancreas therapy as determined for clinical need Starting insulin pump therapy as determined for clinical need On multiple daily injection therapy for insulin delivery

Exclusion Criteria:

* History of ocular disease that may affect the cornea.
* History of corneal trauma or surgery (NB cataract surgery does not preclude enrolment unless surgery occurred in the 3 months prior to enrolment date)
* Concurrent ocular disease, infection or inflammation.
* History of neuropathy due to alcoholism, renal impairment requiring renal replacement therapy, infectious disease (e.g., Lyme disease, HIV/AIDS, hepatitis B), liver failure, B12 deficiency
* Unable to read and comprehend English

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
1. Change in Corneal nerve fibre density (CNFD) | 6 and 12 months
  Corneal nerve fibre density (CNFD)

SECONDARY OUTCOMES:
Neuropathy symptom profile | 6 and 12 months. Min value 0, max value 38. Higher score suggests a worse outcome
  Symptoms of painful neuropathy measured using the neuropathic pain symptom inventory scale
Neuropathy disability score | 6 and 12 months Min value 0, max value 10. Higher score suggests a worse outcome
  Neuropathy disability score
Quality of life questionnaire | 6 and 12 months Min value 0, max value 36. Higher score suggests a worse outcome
  Quality of life Short Form -36 scale measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester Diabetes Centre, Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No